CLINICAL TRIAL: NCT02029196
Title: A Randomised, Parallel Group, Multi-centre Study to Evaluate the Safety Profile of the ITG EVP G1 Product
Brief Title: A Study to Evaluate the Safety Profile of an e-Vapour Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial Brands PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ITG EVP G1 S2
Record Dates: First submitted 2013-12-19; First posted 2014-01-07 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- e-vapour product (EVP) (Experimental): Subjects who switch from using conventional cigarettes to using an e-vapour product (EVP).
  Interventions: Other: E-vapour product
- Conventional cigarette (CC) (Active Comparator): Subjects who continue smoking their usual conventional cigarette (CC) brand.
  Interventions: Other: Conventional cigarette

INTERVENTIONS:
Other: E-vapour product — Smokers of conventional cigarettes who switch to use an e-vapour product.
  Arms: e-vapour product (EVP)
Other: Conventional cigarette — Smokers of conventional cigarettes who continue smoking conventional cigarettes.
  Arms: Conventional cigarette (CC)

SUMMARY:
Electronic Vapour Products (EVPs) is a relatively new class of consumer products that are otherwise known as electronic cigarettes or electronic nicotine delivery devices/systems. These may look like conventional cigarettes but do not contain tobacco.

The 'vapour' produced by such devices typically consists of humectants (propylene glycol or glycerol), nicotine, water, and flavours.

This trial is to evaluate the safety of an e-vapour product.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18-35kg/m2
* Subjects must be established smokers
* Subjects must have smoked five to 30 cigarettes per day for at least one year

Exclusion Criteria:

* Subjects who have used nicotine replacement therapy within 14 days of the screening
* Subjects who have donated blood within 12 months preceding study
* Subjects with relevant illness history
* Subjects positive for hepatitis or Human Immunodeficiency Virus (HIV)
* Subjects with history of drug or alcohol abuse
* Subjects with lung function test or vital signs considered unsuitable
* Subjects who are trying to stop smoking
* Female subjects who are pregnant, or unwilling to use acceptable contraceptive method for the duration of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MD, Principal Investigator — Covance Clinical Research Unit, Springfield House, Hyde Street, Leeds LS2 9LH, UK; Girish Sharma, MD, Principal Investigator — Simbec Research, Merthyr Tydfil, CF48 4DR, UK
Locations (2):
- United Kingdom (2):
  - Covance Clinical Research Unit, Leeds, England
  - Simbec Research, Merthyr Tydfil, Wales

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-vapour Product (EVP) | Conventional Cigarette (CC)
Started | 306 | 102
Completed | 286 | 101
Not Completed | 20 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-vapour Product (EVP) | Conventional Cigarette (CC) | Total
Number analyzed (Participants) | 306 | 102 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.6) | 35.1 (10.6) | 34.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 44 | 182
  Male | 168 | 58 | 226
Exhaled Carbon Monoxide (eCO) [Mean (Standard Deviation); unit: parts per million (ppm)] | 15.8 (6.3) | 16.7 (7.3) | 16.0 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Frequency of adverse events
Time Frame: 12 weeks
Population: All subjects who used the study product at least once.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of adverse events
Arm/Group | E-vapour Product (EVP) | Conventional Cigarette (CC)
Number analyzed (Participants) | 306 | 102
percentage of adverse events | 1.60 [1.55 to 1.65] | 0.79 [0.66 to 0.92]

2. Secondary Outcome: Exhaled Carbon Monoxide
Description: Level of exhaled carbon monoxide at Week 12
Time Frame: 12 weeks
Population: Measure performed on subjects who completed the 12-week study (286 in the e-vapour product arm and 100 in the conventional cigarette arm).
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | E-vapour Product (EVP) | Conventional Cigarette (CC)
Number analyzed (Participants) | 286 | 100
parts per million (ppm) | 8.99 (6.33) | 23.1 (10.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | E-vapour Product (EVP) | Conventional Cigarette (CC)
Serious Adverse Events (participants affected / at risk) | 5/306 | 0/102
Other Adverse Events (participants affected / at risk) | 271/306 | 74/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-vapour Product (EVP) (N=306) | Conventional Cigarette (CC) (N=102)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Puncture wound, left hand, first finger
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Right lobar pneumonia
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) — Sudden death due to severe cardiac arrhythmia as confirmed by post mortem
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-vapour Product (EVP) (N=306) | Conventional Cigarette (CC) (N=102)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 85 (119) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 52 (62) | 8 (9)
Headache (Nervous system disorders) | 145 (372) | 34 (72)
Nasopharyngitis (Infections and infestations) | 34 (36) | 8 (9)
Desire to smoke (Psychiatric disorders) | 84 (86) | 13 (13)
Irritability (General disorders) | 33 (36) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 43 (43) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No